CLINICAL TRIAL: NCT04201197
Title: Interactions Between Cannabinoids and Cytochrome P450-Metabolized Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Washington State University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00207237; U54AT008909 (NIH)
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: Drug-Interactions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo controlled, double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inje Cocktail (Active Comparator): Single oral administration of caffeine (100mg), omeprazole (20mg), losartan (25mg), dextromethorphan (30mg), and midazolam (1mg)
  Interventions: Drug: Inje cocktail
- Inje Cocktail + THC extract (Experimental): Single oral administration of Inje Cocktail + brownie infused with cannabis extract containing 20mg THC
  Interventions: Drug: Inje cocktail; Drug: THC Cannabis extract
- Inje Cocktail + THC/CBD extract (Experimental): Single oral administration of Inje Cocktail + brownie infused with cannabis extract containing 20mg THC and 640mg CBD
  Interventions: Drug: Inje cocktail; Drug: THC/CBD Cannabis Extract

INTERVENTIONS:
Drug: Inje cocktail — Acute drug exposure
Drug: THC Cannabis extract — Acute drug exposure
  Arms: Inje Cocktail + THC extract
Drug: THC/CBD Cannabis Extract — Acute drug exposure
  Arms: Inje Cocktail + THC/CBD extract

SUMMARY:
This study will evaluate drug-drug interactions between cannabis extracts containing Tetrahydrocannabinol (THC) and THC+ Cannabinoids (CBD) and probe drugs for select CYP450 pathways including: caffeine (CYP1A2), omeprazole (CYP2C19), losartan (CYP2C9), dextromethorphan (CYP2D6), and midazolam (CYP3A).

DETAILED DESCRIPTION:
Despite the widespread use and availability of cannabis products, substantive deficiencies remain regarding the potential risks for cannabis or cannabinoids to precipitate adverse interactions with conventional drugs. Evidence from the few systematic clinical studies that have been conducted suggests that THC and CBD can inhibit metabolism of other drugs, via interactions with cytochrome P450 (CYP) enzymes, a large family of enzymes involved in the metabolism of numerous drugs and foreign chemicals in the body. Accordingly, evaluating the potential for drug-drug interactions between cannabis-derived products and common CYP-metabolized drugs merits further investigation. This double-blind, randomized crossover design study will evaluate whether, and to what extent, oral administration of cannabis extracts containing high doses of CBD and/or THC alter the pharmacokinetics of 5 drugs metabolized via CYP pathways including: caffeine (CYP1A2), omeprazole (CYP2C19), losartan (CYP2C9), dextromethorphan (CYP2D6), and midazolam (CYP3A). Healthy adults will complete three experimental dosing sessions, in which participants will orally ingest brownies containing (1) a high THC cannabis extract with a target THC dose of 40mg, (2) a high CBD cannabis extract with a target CBD dose of 1350mg + a THC dose of 40mg, or (3) placebo. In all three experimental dosing sessions, consumption of the cannabis extract infused brownie will be followed by ingestion of a drug "cocktail" comprised of commercial formulations of therapeutic or subtherapeutic doses of each drug. This collection of probe drugs, coined the Inje Cocktail, has been demonstrated to be safe, both administered alone and with various CYP450 inhibitors. At baseline and following administration of the study drugs, a battery of subjective, physiological, and cognitive performance assessments will be completed and biological specimens obtained. Each session will consist of a 12-hour outpatient drug administration visit and a 1-hour outpatient visit the subsequent day for additional biospecimen collection, cognitive testing, and subjective drug effect questionnaires. The study will conclude when 18 participants complete all 3 experimental sessions. The outcomes of this study will be useful to inform clinical decision-making regarding co-administration of cannabinoid-containing products with drugs that are either commonly prescribed by physicians or readily available over-the-counter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult between 18-50 years old
* BMI between 18 to 34 kg/m2
* Willing to use birth control
* Willing to abstain from all medications and citrus fruits for the duration of the study

Exclusion Criteria:

* Medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to drug exposure or completion of other study procedures.
* Use of medications which, in the opinion of the investigator or medical staff, will interfere with the study outcomes or the safety of the participant.
* Clinically significant impairment of kidney, liver, or thyroid function (serum creatinine >1.2 mg/ml (kidney), liver function tests >3x the upper limit of normal (alanine amino transferase >99 U/L; aspartate amino transferase > 99 U/L), and thyroid stimulating hormone > 4.2 uIU/ml), or evidence of current anemia based on blood chemistry testing.
* History of adverse events associated with the ingestion of cannabis or any medications in the Inje cocktail judged by the investigator to present an undue risk of harm to the participant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share protocol information and data to other scientists with reasonable requests for data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the primary outcomes. Availability is indefinite.
Access Criteria: Send request to PI.

REFERENCES:
- [Derived] Zamarripa CA, Spindle TR, Surujunarain R, Weerts EM, Bansal S, Unadkat JD, Paine MF, Vandrey R. Assessment of Orally Administered Delta9-Tetrahydrocannabinol When Coadministered With Cannabidiol on Delta9-Tetrahydrocannabinol Pharmacokinetics and Pharmacodynamics in Healthy Adults: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2254752. doi: 10.1001/jamanetworkopen.2022.54752. PMID 36780161

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a within-subjects design, so all participants were exposed to all three conditions in a randomized order.
Groups:
- Inje Cocktail, Inje Cocktail + THC Extract, Inje Cocktail + THC/CBD Extract: Participants ingested THC, THC/CBD, and the Inje Cocktail in a within-subject crossover design.
Period: Overall Study
Arm/Group | Inje Cocktail, Inje Cocktail + THC Extract, Inje Cocktail + THC/CBD Extract
Started | 22
Placebo, THC, THC+CBD | 3
Placebo, THC+CBD, THC | 3
THC, Placebo, THC+CBD | 3
THC, THC+CBD, Placebo | 3
THC+CBD, THC, Placebo | 3
THC+CBD, THC, Placebo | 3
Completed | 18
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- All Evaluable Study Completers: All study completers completed the following three conditions, in a randomized order:
  1. Single oral administration of Inje Cocktail: caffeine (100mg), omeprazole (20mg), losartan (25mg), dextromethorphan (30mg), and midazolam (1mg)
  2. Single oral administration of Inje Cocktail + brownie infused with cannabis extract containing 20mg THC
  3. Single oral administration of Inje Cocktail + brownie infused with cannabis extract containing 20mg THC and 640mg CBD
Arm/Group | All Evaluable Study Completers
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Losartan Area Under the Curve (AUC) in Plasma
Description: Area under the curve concentration (h*ng/mL) of losartan in plasma using data points obtained 0, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Time Frame: 24 hours
Population: This was a within-subjects design in which all participants were exposed to all three conditions in a randomized order.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Inje Cocktail + Placebo: Single oral administration of Inje Cocktail: caffeine (100mg), omeprazole (20mg), losartan (25mg), dextromethorphan (30mg), and midazolam (1mg)
  + placebo brownie
- Inje Cocktail + THC: Single oral administration of Inje Cocktail + brownie infused with cannabis extract containing 20mg THC
- Inje Cocktail + THC/CBD: Single oral administration of Inje Cocktail + brownie infused with cannabis extract containing 20mg THC and 640mg CBD
Arm/Group | Inje Cocktail + Placebo | Inje Cocktail + THC | Inje Cocktail + THC/CBD
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL | 164 (74) | 185 (72) | 289 (66)

2. Primary Outcome: Peak Change From Baseline Number of Correct Trials on Paced Auditory Serial Addition Task (PASAT)
Description: Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Reported data reflect the peak change from baseline in the total correct trials out of 90 recorded (lower scores indicate worse performance) obtained 1, 2, 3, 4, 6, or 8 hours post-dose.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Correct trials
Arm/Group | Inje Cocktail | Inje Cocktail + THC Extract | Inje Cocktail + THC/CBD Extract
Number analyzed (Participants) | 18 | 18 | 18
Correct trials | -1.1 (14.2) | -6.6 (19.1) | -22.7 (24.6)

3. Primary Outcome: Peak Change From Baseline Cognitive Performance as Assessed by the Divided Attention Task
Description: Cognitive performance will be evaluated with the Divided Attention Task. Reported data reflect the peak change from baseline performance measured as the mean distance (in computer pixels) of the mouse cursor from the central stimulus recorded 1, 2, 3, 4, 6, or 8 hours post-dose. Higher scores indicate worse performance.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Computer pixels
Arm/Group | Inje Cocktail | Inje Cocktail + THC Extract | Inje Cocktail + THC/CBD Extract
Number analyzed (Participants) | 18 | 18 | 18
Computer pixels | -2.1 (9.4) | 15.9 (24.7) | 32.7 (39.2)

4. Primary Outcome: Drug Effect Questionnaire (DEQ) - Peak Score for Feel Drug Effect
Description: The DEQ will be used to obtain subjective ratings of "feel drug effects". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation. Peak rating within 24 hours post-dose is reported.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Inje Cocktail | Inje Cocktail + THC Extract | Inje Cocktail + THC/CBD Extract
Number analyzed (Participants) | 18 | 18 | 18
Score on a scale | 9.4 (27.8) | 59.2 (31.1) | 72.8 (25.9)

5. Primary Outcome: Number of Correct Trials on the Digit Symbol Substitution Task (DSST)
Description: Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Results reported reflect the peak change from baseline on the total correct trials in 90 seconds (lower scores indicate worse performance) assessed 1, 2, 3, 4, 6, or 8 hours post-dose.
Time Frame: 8 hours
Population: All participants were exposed to each of the 3 conditions
Measure: Mean (Standard Deviation); unit: Correct trials
Arm/Group | Inje Cocktail | Inje Cocktail + THC Extract | Inje Cocktail + THC/CBD Extract
Number analyzed (Participants) | 18 | 18 | 18
Correct trials | 2.5 (7.5) | -2.7 (11.2) | -9.9 (17.6)

6. Primary Outcome: Peak Change From Baseline Beats Per Minute for Heart Rate (HR)
Description: HR will be obtained using an automated monitor to evaluate changes in beats per minute as a function of conditions. Data reflect the peak change from baseline measured 1, 2, 3, 4, 6, or 8 hours post-dose.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Inje Cocktail | Inje Cocktail + THC Extract | Inje Cocktail + THC/CBD Extract
Number analyzed (Participants) | 18 | 18 | 18
Beats per minute | -4.4 (12.4) | 10.1 (14.1) | 25.4 (20.9)

7. Secondary Outcome: Caffeine AUC in Plasma
Description: Area under the curve concentration (h*ng/mL) of caffeine in plasma using data points obtained 0, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Time Frame: 24 hours
Population: This was a within-subjects design in which all participants were exposed to all three conditions in a randomized order.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Inje Cocktail + Placebo | Inje Cocktail + THC | Inje Cocktail + THC/CBD
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL | 18948 (58) | 18554 (61) | 26264 (56)

8. Secondary Outcome: Omeprazole AUC in Plasma
Description: Area under the curve concentration (h*ng/mL) of omeprazole in plasma using data points obtained 0, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Time Frame: 24 hours
Population: This was a within-subjects design in which all participants were exposed to all three conditions in a randomized order.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Inje Cocktail + Placebo | Inje Cocktail + THC | Inje Cocktail + THC/CBD
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL | 385 (90) | 379 (86) | 1183 (86)

9. Secondary Outcome: Dextromethorphan AUC in Plasma
Description: Area under the curve concentration (h*ng/mL) of dextromethorphan in plasma using data points obtained 0, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Time Frame: 24 hours
Population: This was a within-subjects design in which all participants were exposed to all three conditions in a randomized order.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Inje Cocktail + Placebo | Inje Cocktail + THC | Inje Cocktail + THC/CBD
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL | 10.4 (108) | 13.2 (112) | 13.6 (104)

10. Secondary Outcome: Midazolam AUC in Plasma
Description: Area under the curve concentration (h*ng/mL) of midazolam in plasma using data points obtained 0, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Time Frame: 24 hours
Population: This was a within-subjects design in which all participants were exposed to all three conditions in a randomized order.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Inje Cocktail + Placebo | Inje Cocktail + THC | Inje Cocktail + THC/CBD
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL | 23 (101) | 24 (75) | 36 (84)

ADVERSE EVENTS:
Time Frame: up to 38 days
Groups:
- Inje Cocktail + Placebo: Participants ingested the Inje Cocktail and a brownie containing no cannabis
- Inje Cocktail + THC: Participants ingested the Inje Cocktail and a brownie containing 20mg THC
- Inje Cocktail + THC+CBD: Participants ingested the Inje Cocktail and a brownie containing 20mg THC and 640mg CBD
Arm/Group | Inje Cocktail + Placebo | Inje Cocktail + THC | Inje Cocktail + THC+CBD
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 8/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inje Cocktail + Placebo (N=22) | Inje Cocktail + THC (N=22) | Inje Cocktail + THC+CBD (N=22)
Nausea (Gastrointestinal disorders) | 0 | 0 | 6 (6)
Emesis (Gastrointestinal disorders) | 0 | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04201197/Prot_SAP_000.pdf